CLINICAL TRIAL: NCT01921816
Title: A Study on the Efficacy and Safety of Continuous Renal Replacement Therapy (CVVHDF) Using a Commercial Citrate-containing Replacement Fluid (Prismocitrate 18/0)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lui Mei Sze, Doctor, Queen Mary Hospital, Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UW 12-173
Record Dates: First submitted 2013-07-31; First posted 2013-08-13 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency

ARMS (1):
- Prismocitrate 18/0 (Other): citrate-containing replacement solution (Prismocitrate 18/0, Gambro) will be administered at pre-filter port during continuous hemodiafiltration, for the purpose as replacement solution and anticoagulation
  Interventions: Device: Prismocitrate 18/0, Prism0cal

INTERVENTIONS:
Device: Prismocitrate 18/0, Prism0cal — Subjects on continuous hemodiafiltration will ordinarily receive heparin as the anticoagulation. In our study, regional citrate anticoagulation with Prismacitrate is used to replace heparin. Citrate has been shown in study to be safer than heparin with reduced bleeding risk
  Other Names: Prismocitrate 18/0 (replacement solution), Prism0cal (dialysate), Gambro

SUMMARY:
The investigators aim to examine the efficacy and safety of using a new citrate containing commercially available solutions (Prismocitrate 18/0) as the regional citrate anticoagulation in continuous renal replacement therapy for critically ill patients.

DETAILED DESCRIPTION:
Acute kidney injury is common in critically ill patients, and continuous renal replacement therapy is the preferable mode of treatment to remove the metabolic waste while avoiding the hemodynamic instability associated with intermittent hemodialysis. Thrombosis frequently occurs in the hemofilter which could reduce the circuit lifespan, jeopardize the efficacy of renal replacement, result in loss of blood cells and increased transfusion requirement. Anticoagulants including conventional heparin and low molecular weight heparin, introduced via the arterial port of the circuit, are widely used to reduce clotting within the extracorporeal circuit. However, significant amount of heparin is not removed in the circuit and will be carried into patient's circulation, which could lead to bleeding complications. Regional citrate anticoagulation (RCA) has been used for intermittent haemodialysis since 1983, and its use has extended to that for continuous renal replacement therapy (CRRT) since 1987. Citrate is introduced at therapeutic level at the arterial limb of the dialysis circuit, where it chelates calcium ions in the blood to prevent clotting within the hemofilter. While some calcium-citrate complex is removed in the filter, the residual will be circulated to the patient and be metabolized in liver. Patient's systemic ionized calcium level remains normal, by hemodilution and also calcium replacement. Therefore, the anticoagulant effect from citrate is regional and confined to the extracorporeal circuit. RCA has the potential to extend circuit life during renal replacement therapy without systemic anticoagulation. In a recent meta-analysis of randomized controlled trials, RCA was as efficacious as heparin anticoagulation in term of maintaining circuit function, and RCA was associated with decreased risk of bleeding with no significant increase in incidence of metabolic alkalosis.(5) Hypocalcemia was more common in patients receiving citrate, but of note, no clinical adverse event was reported in the included studies. Although citrate anticoagulation had repeatedly been demonstrated to prolong filter life, many hospitals still refrained from using it, as a result of limited experience, different patient variety, or other reasons.

The investigators' group has performed a pilot study (HKU/HA HKW IRB No: UW 08-221) to assess the efficacy and safety of continuous venous-venous hemodiafiltration(CVVHDF) using a commercial citrate containing replacement fluid (Prismocitrate 10/2, Gambro) which contains 10mmol/l citrate and 2 mmol/l citric acid. 15 subjects were recruited from July 2008 to June 2011. No serious adverse events were reported, including severe hypocalcemia, hypercalcemia, citrate toxicity and severe acid base disturbances. Metabolic acidosis due to renal failure were only partially corrected by CRRT with citrate anticoagulation in the initial study subjects, the problem was subsequently solved by adding supplemental bicarbonate to the dialysate. Since then, all the patients were able to complete the treatment protocols with adequate kidney lifespan, correction of metabolic abnormalities and fluid imbalance. However, since additional bicarbonate is needed to correct the metabolic acidosis during CRRT, there is room for improvement regarding the formulation of the citrate-containing solution to reduce acid liberation while increasing the alkali bicarbonate production. Prismocitrate 18/0, which contains 18mmol/l citrate (one mmol citrate could be metabolized to produce 3 mmol bicarbonate) and no citric acid, could potentially result in better acid-base control during CRRT.

ELIGIBILITY:
Inclusion Criteria:

* The patient requires CRRT as treatment for renal failure, as decided by the attending physician
* The patient fulfils at least one of the following clinical criteria for initiating CRRT:

  1. According to the RIFLE criteria, (11) patients satisfying the "injury" criteria (increase creatinine by 2 fold or urine output<0.5ml/kg/hr for 12hr) will be considered for CRRT
  2. Hyperkalemia ([K+] > 6.5 mmol/L).
  3. Severe acidemia (pH < 7.2).
  4. Urea > 25 mmol/liter.
  5. Clinically significant organ oedema in the setting of ARF.

     Exclusion Criteria:

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
filter lifespan | up to 4 days
  filter lifespan will be recorded as the time duration from commencement of renal replacement therapy till filter clotted or therapy ended

SECONDARY OUTCOMES:
metabolic and electrolyte control | up to 4days
  Serum electrolytes (calcium, sodium, potassium, magnesium, acid-base)will be monitored at baseline, then every 6 hours onwards during the CRRT
bleeding/transfusion requirement | up to 4 days
  blood counts including the hemoglobin level and patient clinical status will be monitored at baseline, then once everyday during renal replacement therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Adult Intensive Care unit, Queen Mary Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Background] Oudemans-van Straaten HM, Kellum JA, Bellomo R. Clinical review: anticoagulation for continuous renal replacement therapy--heparin or citrate? Crit Care. 2011 Jan 24;15(1):202. doi: 10.1186/cc9358. PMID 21345279
- [Background] Leung AK, Shum HP, Chan KC, Chan SC, Lai KY, Yan WW. A retrospective review of the use of regional citrate anticoagulation in continuous venovenous hemofiltration for critically ill patients. Crit Care Res Pract. 2013;2013:349512. doi: 10.1155/2013/349512. Epub 2013 Jan 28. PMID 23424680
- [Background] Shum HP, Chan KC, Yan WW. Regional citrate anticoagulation in predilution continuous venovenous hemofiltration using prismocitrate 10/2 solution. Ther Apher Dial. 2012 Feb;16(1):81-6. doi: 10.1111/j.1744-9987.2011.01001.x. Epub 2011 Oct 3. PMID 22248200